CLINICAL TRIAL: NCT04793880
Title: Integrating Cost Into Shared Decision-Making for Heart Failure With Reduced Ejection Fraction
Brief Title: Cost and Shared Decision-Making for Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Neal Dickert, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002215; 1R01HS026081-01 (AHRQ)
Record Dates: First submitted 2021-02-23; First posted 2021-03-11 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Chronic Heart Failure
Keywords: Out-of-pocket cost; Shared decision-making; Heart failure with reduced ejection fraction (HFrEF)

STUDY DESIGN:
Intervention Model Description: This study utilizes a stepped wedge cluster-randomized design where study sites are assigned to transition to the intervention as recruitment milestone are met.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medication checklist with cost information (Experimental): Participants with chronic heart failure with reduced ejection fraction (HFrEF) having a clinic visit at a site randomized to the medication checklist with cost information intervention.
  Interventions: Behavioral: Medication Cost Information; Behavioral: Heart Failure Medicines Checklist
- Medication checklist (Active Comparator): Participants with chronic heart failure with reduced ejection fraction (HFrEF) having a clinic visit at a site randomized to the medication checklist without cost information.
  Interventions: Behavioral: Heart Failure Medicines Checklist

INTERVENTIONS:
Behavioral: Medication Cost Information — This version of the HFrEF medication checklist includes patient-specific estimated monthly out-of-pocket cost for each medication. TailorMed, a company designed to provide financial counseling and planning for patients, will generate the patients' out-of-pocket cost based on insurance status. The costs for non-generic HFrEF medications will then be populated onto a checklist of recommended heart failure medications so that patients and their clinicians will have this information available during their clinical encounter.
  Arms: Medication checklist with cost information
Behavioral: Heart Failure Medicines Checklist — The Heart Failure Medicines Checklist is an evidence-based medication checklist that describes guideline-recommended medications for HFrEF. This tool is used during the clinical encounter to facilitate a discussion about medications that may be most appropriate for the patient.

SUMMARY:
This study is designed to understand the impact of providing patient-specific cost at the time of the clinical encounter on decision-making for heart failure medications. The researchers will provide patients with heart failure with patient-specific cost information for non-generic heart failure medications. This cost information will be populated onto a checklist of recommended HF medications so that patients and their clinicians will have this information available during their clinical encounter. Patients in the control arm will receive the same checklist but without the cost information.

DETAILED DESCRIPTION:
For many years, medical treatment of heart failure with reduced ejection fraction (HFrEF) was defined by a combination of low-cost, generic medications. Recently, new medications have demonstrated reductions in mortality and hospitalization. These include the angiotensin receptor blocker and neprilysin inhibitor (ARNI) sacubitril-valsartan, sodium-glucose cotransporter-2 inhibitors (SGLT2I), and ivabradine. These medications all carry important clinical benefits but also are more expensive, with co-payments varying significantly but often in the range of $50-$100 per month. These costs are highly relevant for patients' decisions, especially for patients who have Medicare Part D drug coverage and are not eligible for co-pay assistance programs.

Prior research has demonstrated that patients are sensitive to costs regarding HFrEF medications and receptive to cost discussions with clinicians. Some broad efforts at price transparency have been promoted, but generic price information is of little value to patients and clinicians when out-of-pocket costs vary significantly from patient to patient based on insurance coverage. At present, neither clinicians nor patients have out-of-pocket costs available at the time of clinical encounters in order to facilitate integration of this information into decisions.

The objective of this trial is to examine the impact of integrating patient-specific out-of-pocket cost into shared decision-making regarding heart failure medications in patients with HFrEF. This will be performed by integrating patient-specific cost into an existing, evidence-based checklist for HFrEF medications. The study will utilize a simple cluster-randomized design. All patients in the study will receive, at the time of a clinical encounter, an evidence-based heart failure medication checklist that describes guideline-recommended medications for HFrEF. Patients in the intervention group will receive a version of the checklist that also includes their estimated co-payment for non-generic heart failure medications based upon their insurance status at the time of the encounter.

This study is designed as a preliminary trial to understand the real impact of providing patient-specific cost at the time of the clinical encounter. The researchers will audio record clinical encounters, conduct a follow-up survey with participants, and collect follow-up data regarding each patient's medications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HFrEF (ejection fraction < 40%)
* Outpatient clinical encounter with cardiologist (virtual or in-person)

Exclusion Criteria:

* Advanced HF therapy (LVAD or transplant or undergoing active workup or listing for these therapies; home inotrope usage)
* Patient currently in hospice care or with known life expectancy under 1 year
* Dialysis-dependence or glomerular filtration rate (GFR) < 30 (due to medication contraindications)
* Pregnancy (because many guideline-recommended drugs, including those with associated high costs, are not approved for use in pregnancy)
* Non-English speaking (because of the absence of non-English speaking research staff to communicate with non-English speaking patients and to qualitatively analyze/code audio-recorded data)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Discussed Medication Cost | Day 1 (during clinic encounter)
  The number of patients whose clinic encounters involved a discussion of heart failure medication cost will be compared between study arms. The discussion of heart failure medication cost is a binary outcome of whether or not the cost of heart failure medication was discussed during the recorded clinical encounter. Any mention of heart failure medication cost will be counted as a cost discussion. The primary outcome will be analyzed using a generalized linear mixed model, with covariates including clinic site, time, age, race, sex, insurance status, and income. Potentially different intervention effects by site and patient characteristics will be examined.

SECONDARY OUTCOMES:
Physician Recommendation Coding System (PhyReCS) Score | Day 1 (during clinic encounter)
  The strength of the clinical recommendation for a medication will be assessed with the Physician Recommendation Coding System (PhyReCS) scale, using the audio recording of the clinic encounter. The PhyReCS is a 5-point scale indicating how strongly the physician recommended a particular treatment. A strong recommendation is coded as +2, a mild recommendation is +1, recommendations neither for nor against treatment are coded as 0, a mild recommendation against treatment is -1, and a strong recommendation against treatment is coded as -2.
Length of discussion | Day 1 (during clinic encounter)
  The length of medication cost discussion will be measured in minutes, using the audio recording of the clinic encounter.
Helpfulness of medication checklist score | 2 to 3 weeks after clinic encounter
  Participants will rate how helpful they found the medication checklist to be on a 5-point scale where 1 = extremely helpful and 5 = not helpful at all.
Helpfulness of medication checklist with price information score | 2 to 3 weeks after clinic encounter
  Participants in the intervention arm will rate how helpful they found the price information included on the medication checklist to be on a 5-point scale where 1 = extremely helpful and 5 = not helpful at all.
Low Literacy Decisional Conflict Scale score | 2 to 3 weeks after clinic encounter
  Participant perception of the visit with their doctor will be assessed with the Low Literacy Decisional Conflict Scale (DCS). The DCS includes 10 questions which are responded to as yes (scored as 0), no (scored as 4), or unsure (scored as 2). Total scores range from 0 to 40 with low scores indicating less difficulty in understanding treatment options.
Consumer Assessment of Healthcare Providers and Systems (CAHPS®) Clinician & Group Survey score | 2 to 3 weeks after clinic encounter
  To assess participant perceptions of their doctor, questions 14-18 of the CAHPS Clinician & Group Survey - Adult Visit 4.0 (beta) instrument will be used. Responses are given on a 3-point scale where 1 = yes, definitely, 2 = yes, somewhat, and 3 = no. The total score of these 4 items range from 4 to 12 with lower scores indicating a more positive experience with their healthcare provider.
Prescription of non-generic medications | Day 1 (during clinic encounter)
  The number of participants prescribed non-generic medications at the clinic encounter will be obtained from electronic medical records.
Medication persistence | 3 months after clinic encounter
  The number of participants continuing to take their prescribed medication three months after the clinic encounter will be obtained from electronic medical records.
Clinician perceptions | End of study (up to 26 months)
  Clinician perceptions will be assessed qualitatively through focus group interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Neal W Dickert, MD, PhD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - UCHealth Heart and Vascular Center Clinics, Aurora, Colorado
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Emory University Hospital, Atlanta, Georgia
  - Emory St. Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available for sharing upon request, including survey data, electronic health record data, and transcribed interviews.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available one year after publication of the main results.
Access Criteria: Data will be available for sharing with investigators seeking to verify analyses or to conduct additional analyses that are appropriate to the nature of these data. Data will be made available for sharing upon request, after execution of a data sharing agreement.

REFERENCES:
- [Derived] Dickert NW, Speight CD, Balser M, Biermann H, Davis JK, Halpern SD, Ko YA, Krishnan A, Matlock DD, Mitchell AR, Moore MA, Montembeau SC, Morris AA, Noonan K, Rao BR, Scherer LD, Sloan CE, Ubel PA, Allen LA. Integrating Out-of-Pocket Costs Into Shared Decision-Making for Heart Failure With Reduced Ejection Fraction: A Stepped-Wedge Trial (POCKET-COST-HF). Circ Cardiovasc Qual Outcomes. 2025 Jan;18(1):e011273. doi: 10.1161/CIRCOUTCOMES.124.011273. Epub 2024 Dec 3. PMID 39624892
- [Derived] Montembeau SC, Rao BR, Mitchell AR, Speight CD, Allen LA, Halpern SD, Ko YA, Matlock DD, Moore MA, Morris AA, Scherer LD, Ubel P, Dickert NW. Integrating Cost into Shared Decision-Making for Heart Failure with Reduced Ejection Fraction (POCKET-COST-HF): A Trial Providing Out-of-Pocket Costs for Heart Failure Medications during Clinical Encounters. Am Heart J. 2024 Mar;269:84-93. doi: 10.1016/j.ahj.2023.11.013. Epub 2023 Dec 12. PMID 38096946

DOCUMENTS (1):
  • Informed Consent Form (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT04793880/ICF_000.pdf